CLINICAL TRIAL: NCT00836459
Title: A Randomised Controlled Trial and Cost-effectiveness Evaluation of "Booster" Interventions to Sustain Increases in Physical Activity in Middle-aged Adults in Deprived Urban Neighbourhoods.
Brief Title: Sheffield Physical Activity Booster Trial
Acronym: Booster
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Richard Hudson (Other)
Collaborators: NHS Health Technology Assessment Programme (Other)
Responsible Party: Sponsor-Investigator, Richard Hudson, Sponsor, University of Sheffield
Organization: University of Sheffield (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 120243; HTA: 07/25/02; IRAS: 08/H1308/270
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Public Health
Keywords: Humans; Middle Aged; Behavior Therapy; Directive Counseling; Health Behavior; Interview, Psychological; Motivation; Exercise; Physical Fitness; Self Efficacy; Life Style; Health Promotion; Health Knowledge, Attitudes, Practice; Body Mass Index; Monitoring, Ambulatory; Walking
MeSH Terms: conditions — Health Behavior; Motor Activity; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention)
- Mini Booster (Experimental)
  Interventions: Behavioral: Mini Booster
- Full Booster (Experimental)
  Interventions: Behavioral: Full Booster

INTERVENTIONS:
Behavioral: Mini Booster — Two telephone-based physical activity consultations, delivered in a motivational interviewing style, at one month and two months from randomisation
  Arms: Mini Booster
Behavioral: Full Booster — Two face-to-face physical activity consultations, delivered in a motivational interviewing style, at one month and two months from randomisation
  Arms: Full Booster

SUMMARY:
Adults that increase their physical activity can improve their health, and reduce future risks to health, but long-term changes are difficult to sustain. This study assesses whether it is worth providing further support, 3 months after giving initial advice, to those who have managed to do more physical activity. All participants will initially be given an interactive DVD. A researcher from Sheffield Hallam University will provide two telephone follow ups at one month intervals to assess physical activity levels. Only those that have increased their physical activity at this point will remain in the study. These participants will receive a "mini booster", a "full booster" or no booster. The "mini booster" consists of a two telephone calls one month apart to discuss physical activity and usage of the DVD. A "full booster" consists of a face-to-face meeting with the facilitator at the same intervals. The purpose of these booster sessions is to help the individual to maintain their increase in physical activity. The investigators will measure the differences in physical activity, quality of life and costs, associated with the booster interventions, 3 months and 9 months from randomisation. The research will be carried out in 20 of the most deprived neighbourhoods in Sheffield. These locations have large, ethnically diverse populations, high levels of economic deprivation, low levels of physical activity, poorer health and shorter life expectancy. Participants will be recruited through general practices and community groups, as well as by postal invitation to ensure the participation of minority ethnic groups and those with lower levels of literacy. Sheffield City Council and Primary Care Trust fund a range of facilities and activities to promote physical activity and variations in access to these between neighbourhoods will make it possible to examine whether the effectiveness of the intervention is modified by access to community facilities.

ELIGIBILITY:
Inclusion Criteria:

* Residents of the 20 most deprived neighbourhoods in the city of Sheffield
* Aged 40 to 64 years
* Not achieving the current recommended activity level (30 mins of moderate activity on at least 5 days) assessed using the SPAQ (Lowther, 1999) and wishing to have support to become more active

Exclusion Criteria:

* Have increased their physical activity level by at least 30 mins of moderate or vigorous activity per week (assessed using the SPAQ) since initial assessment of activity level
* Capacity to give written informed consent to trial participation

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 282 (Actual)
Dates: Start 2009-11; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Physical activity measured by accelerometry. | 3 months post-randomisation

SECONDARY OUTCOMES:
Physical activity assessed by accelerometry. | 9 months post-randomisation
Self-reported moderate or strenuous physical activity using the Scottish Physical Activity Questionnaire (SPAQ, incorporating Stage of Change information) which records type and duration of activities in the previous week | 3 months and 9 months post-randomisation
Health-related quality of life using the Sheffield Version SF-12v2 plus 4 survey instrument | 3 months and 9 months post-randomisation
Self-reported use of community facilities for physical activity | 3 months and 9 months post-randomisation
Self-reported health and social care contacts | 3 months and 9 months post-randomisation
Psychological measures of motivation, assessed using BREQ-2 (Mullan et al, 1997) | 3 months and 9 months post-randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Liddy Goyder, MD FFPH, Principal Investigator — University of Sheffield
Locations (1):
- Centre for Sport and Exercise Science, Sheffield Hallam University, Sheffield, South Yorkshire, United Kingdom

REFERENCES:
- [Result] Goyder, Elizabeth, et al.
- [Derived] Copeland RJ, Horspool K, Humphreys L, Scott E; Booster trial team. Recruiting to a large-scale physical activity randomised controlled trial - experiences with the gift of hindsight. Trials. 2016 Feb 24;17(1):104. doi: 10.1186/s13063-016-1229-0. PMID 26908117
- [Derived] Goyder E, Hind D, Breckon J, Dimairo M, Minton J, Everson-Hock E, Read S, Copeland R, Crank H, Horspool K, Humphreys L, Hutchison A, Kesterton S, Latimer N, Scott E, Swaile P, Walters SJ, Wood R, Collins K, Cooper C. A randomised controlled trial and cost-effectiveness evaluation of 'booster' interventions to sustain increases in physical activity in middle-aged adults in deprived urban neighbourhoods. Health Technol Assess. 2014 Feb;18(13):1-210. doi: 10.3310/hta18130. PMID 24571932
- [Derived] Hind D, Scott EJ, Copeland R, Breckon JD, Crank H, Walters SJ, Brazier JE, Nicholl J, Cooper C, Goyder E. A randomised controlled trial and cost-effectiveness evaluation of "booster" interventions to sustain increases in physical activity in middle-aged adults in deprived urban neighbourhoods. BMC Public Health. 2010 Jan 4;10:3. doi: 10.1186/1471-2458-10-3. PMID 20047672